CLINICAL TRIAL: NCT06303726
Title: Comparison of Single-bundle Versus Double-bundle Anterior Cruciate Ligament Reconstruction: Short-term and Long-term Function and Imaging Results
Brief Title: Comparison of Single-bundle Versus Double-bundle Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRP-2021/02-19
Record Dates: First submitted 2023-07-27; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-07

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: anterior cruciate ligament; bone to bone (BTB); single bundle; double bundle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single bundle ACL reconstruction (Active Comparator): In this group we chose to do surgery of ACL reconstruction with single bundle (patellar ligament).
  Interventions: Procedure: ACL reconstruction single bundle
- Double bundle ACL reconstruction (Active Comparator): In this group we chose to do surgery of ACL reconstruction with double bundle - hamstring ligament.
  Interventions: Procedure: ACL reconstruction double bundle

INTERVENTIONS:
Procedure: ACL reconstruction single bundle — We will do surgery of ACL reconstruction with patellar ligament.
  Arms: Single bundle ACL reconstruction
Procedure: ACL reconstruction double bundle — We will do surgery of ACL reconstruction with hamstring ligament.
  Arms: Double bundle ACL reconstruction

SUMMARY:
The goal of this retrospective randomized study is to compare two surgical techniques (single vs. double bundle) of ACL (anterior cruciate ligament) reconstructions in participants with rupture of anterior cruciate ligament without major other injuries of the injured knee (exclusion criteria defined).

The main question it aims to answer are:

* which surgery gives better outcome in patients (short- and long-term results)?
* are there any sings of osteoarthritis in an injured knee compared to a healthy knee?

Participants will be invited to our clinic after 15 years to do clinical and functional exams with x-Ray and magnetic resonance imaging (MRI) of both knees. Subjective exams with different scores (Tegner score, Lysholm score..) were also done. The same exam protocol for participant was used again after two years and fifteen years since surgery.

DETAILED DESCRIPTION:
Double bundle (DB) ACL reconstruction has gained popularity in the last few years. Biomechanical and intra - operative studies have shown better antero - posterior and rotational stability after DB vs. single bundle (SB) reconstruction. However, only few studies are found in the literature that have evaluated and compared clinical results between SB and DB ACL reconstruction. All reported studies used hamstrings in both DB and SB techniques. No studies were found that used patellar tendon autograft for the SB.

The purpose of the present study was therefore to evaluate and compare the clinical results of DB hamstring and SB patellar tendon ACL reconstruction techniques.

A total of 40 patients (29 male and 11 female, average (SD) age 36) were randomized during routine surgery (2 years after the surgery) into either double bundle (DB) or single bundle (SB) group. Patients with combined (medial, lateral or posterior) ligamentous injuries were not included in the study. ACL reconstruction in DB group was done by four tunnel hamstring technique with EndoButton femoral and cancellous screw tibial fixation. In the SB group patellar tendon autograft was fixed with titanium interference screws. The same postoperative rehabilitation protocols were used for both groups.

Subjective evaluation comprised IKDC (International Knee Documentation Committee) subjective score, Tegner activity and Lysholm scores. Objective evaluation was done by the IKDC 2000 knee examination protocol. Antero - posterior stability was measured by KT 2000 (knee arthrometer) and by Rollimeter. One leg hop test was performed to assess the functional results. Isokinetic thigh muscle strength measurements on Biodex isokinetic dynamometer were performed.

The same protocol was performed for the clinical exams after 15 years since surgery. A total of 30 patients were examen. Investigators also did imaging of both knees (X-ray and MRI) for checking the sings of osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* complete ACL rupture
* symptoms and clinical sings for rupture of ACL (instability of knee, swelling, pain, reduced knee function,...)
* patient consent
* magnetic resonance with this of kind injury

Exclusion Criteria:

* associated injuries to other knee ligaments
* major meniscus injuries
* X-ray abnormalities of injured knee
* preliminary ACL reconstruction
* associated injury to the other knee

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
IKDC SUBJECTIVE SCORE | before surgery, 2 years and 15 years after surgery
  Daily activities, limitations
TEGNER SCORE | 2 years and 15 years after surgery
  Daily activities, limitations
LYSHOLM SCORE | 2 years and 15 years after surgery
  Daily activities, limitations
OBJECTIVE PARAMETER: STREENGHT OF FLEXORS AND EXTENSORS | 2 years and 15 years after surgery
  Measurements with Biodex isokinetic Dynamometer (deficit (%) at 60 deg/s and 180 deg/s; operated to nonoperated ratio (total work))
OBJECTIVE PARAMETER: AP TRANSLATION (anterior-posterior) | 2 years and 15 years after surgery
  Measured by KT 1000 and Rollimeter. Laxity was expressed as the difference between injured knee and uninjured knee in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Kozic, Study Chair — University Clinical Center Maribor
Locations (1):
- University Clinical Center Maribor, Maribor, Slovenia

IPD SHARING:
Plan to Share IPD: No
Fo now we are not planning to share any participant data to other researchers.

REFERENCES:
- [Background] Maynard MJ, Deng X, Wickiewicz TL, Warren RF. The popliteofibular ligament. Rediscovery of a key element in posterolateral stability. Am J Sports Med. 1996 May-Jun;24(3):311-6. doi: 10.1177/036354659602400311. PMID 8734881
- [Background] Freeman MA, Pinskerova V. The movement of the knee studied by magnetic resonance imaging. Clin Orthop Relat Res. 2003 May;(410):35-43. doi: 10.1097/01.blo.0000063598.67412.0d. PMID 12771815
- [Background] Browne C, Hermida JC, Bergula A, Colwell CW Jr, D'Lima DD. Patellofemoral forces after total knee arthroplasty: effect of extensor moment arm. Knee. 2005 Apr;12(2):81-8. doi: 10.1016/j.knee.2004.05.006. PMID 15749440
- [Background] Nuno N, Ahmed AM. Sagittal profile of the femoral condyles and its application to femorotibial contact analysis. J Biomech Eng. 2001 Feb;123(1):18-26. doi: 10.1115/1.1339819. PMID 11277297
- [Background] Siu D, Rudan J, Wevers HW, Griffiths P. Femoral articular shape and geometry. A three-dimensional computerized analysis of the knee. J Arthroplasty. 1996 Feb;11(2):166-73. doi: 10.1016/s0883-5403(05)80012-9. PMID 8648311
- [Background] Lonner JH, Jasko JG, Thomas BS. Anthropomorphic differences between the distal femora of men and women. Clin Orthop Relat Res. 2008 Nov;466(11):2724-9. doi: 10.1007/s11999-008-0415-0. Epub 2008 Aug 22. PMID 18719975
- [Background] Griffin FM, Insall JN, Scuderi GR. The posterior condylar angle in osteoarthritic knees. J Arthroplasty. 1998 Oct;13(7):812-5. doi: 10.1016/s0883-5403(98)90036-5. PMID 9802670
- [Background] Yoon KH, Kim JS, Kim SJ, Park M, Park SY, Park SE. Eight-year results of transtibial nonanatomic single-bundle versus double-bundle anterior cruciate ligament reconstruction: Clinical, radiologic outcomes and survivorship. J Orthop Surg (Hong Kong). 2019 May-Aug;27(2):2309499019840827. doi: 10.1177/2309499019840827. PMID 30955412
- [Background] Freedman KB, D'Amato MJ, Nedeff DD, Kaz A, Bach BR Jr. Arthroscopic anterior cruciate ligament reconstruction: a metaanalysis comparing patellar tendon and hamstring tendon autografts. Am J Sports Med. 2003 Jan-Feb;31(1):2-11. doi: 10.1177/03635465030310011501. PMID 12531750
- [Background] Adravanti P, Dini F, de Girolamo L, Cattani M, Rosa MA. Single-Bundle versus Double-Bundle Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Controlled Trial with 6-Year Follow-up. J Knee Surg. 2017 Nov;30(9):898-904. doi: 10.1055/s-0037-1598176. Epub 2017 Feb 20. PMID 28219088
- [Background] Hefti F, Muller W, Jakob RP, Staubli HU. Evaluation of knee ligament injuries with the IKDC form. Knee Surg Sports Traumatol Arthrosc. 1993;1(3-4):226-34. doi: 10.1007/BF01560215. PMID 8536037
- [Background] Shaieb MD, Kan DM, Chang SK, Marumoto JM, Richardson AB. A prospective randomized comparison of patellar tendon versus semitendinosus and gracilis tendon autografts for anterior cruciate ligament reconstruction. Am J Sports Med. 2002 Mar-Apr;30(2):214-20. doi: 10.1177/03635465020300021201. PMID 11912091
- [Background] Jarvela S, Kiekara T, Suomalainen P, Jarvela T. Double-Bundle Versus Single-Bundle Anterior Cruciate Ligament Reconstruction: A Prospective Randomized Study With 10-Year Results. Am J Sports Med. 2017 Sep;45(11):2578-2585. doi: 10.1177/0363546517712231. Epub 2017 Jun 29. PMID 28661696
- [Background] Briggs KK, Steadman JR, Hay CJ, Hines SL. Lysholm score and Tegner activity level in individuals with normal knees. Am J Sports Med. 2009 May;37(5):898-901. doi: 10.1177/0363546508330149. Epub 2009 Mar 23. PMID 19307332
- [Background] Marmura H, Getgood AMJ, Spindler KP, Kattan MW, Briskin I, Bryant DM. Validation of a Risk Calculator to Personalize Graft Choice and Reduce Rupture Rates for Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2021 Jun;49(7):1777-1785. doi: 10.1177/03635465211010798. Epub 2021 May 4. PMID 33945339